CLINICAL TRIAL: NCT06660654
Title: REJOICE-PanTumor01: A Phase 2, Multicenter, Open-Label, Pan-Tumor Trial to Evaluate Efficacy and Safety of Raludotatug Deruxtecan (R-DXd) in Participants With Advanced/Metastatic Solid Tumors
Brief Title: A Study of Raludotatug Deruxtecan in Participants With Advanced/Metastatic Solid Tumors (REJOICE-PanTumor01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS6000-126; 2024-513307-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumors
Keywords: Advanced/metastatic solid tumors; Raludotatug Deruxtecan; R-DXd; DS-6000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Endometrial Cancer Cohort (Experimental): Participants with endometrial cancer who will receive raludotatug deruxtecan (R-DXd) administered intravenously every 3 weeks (Q3W).
  Interventions: Drug: Raludotatug deruxtecan
- Cervical Cancer Cohort (Experimental): Participants with cervical cancer who will receive R-DXd administered intravenously Q3W.
  Interventions: Drug: Raludotatug deruxtecan
- Non-high-grade Serous Ovarian Cancer (Experimental): Participants with non-high-grade serous ovarian cancer who will receive R-DXd administered intravenously Q3W.
  Interventions: Drug: Raludotatug deruxtecan
- Urothelial Cancer Cohort (Experimental): Participants with urothelial cancer who will receive R-DXd administered intravenously Q3W.
  Interventions: Drug: Raludotatug deruxtecan
- Clear Cell Renal Carcinoma (ccRCC) Cohort (Experimental): Participants with clear cell renal carcinoma (ccRCC) who will receive R-DXd administered intravenously Q3W.
  Interventions: Drug: Raludotatug deruxtecan

INTERVENTIONS:
Drug: Raludotatug deruxtecan — IV administration Q3W
  Other Names: R-DXd

SUMMARY:
This pan-tumor trial is designed as a signal-seeking trial to assess efficacy and safety of raludotatug deruxtecan (R-DXd) monotherapy in locally advanced or metastatic solid tumors with various cadherin-6 (CDH6) expression levels, including gynecological cancers (endometrial cancer, cervical cancer, and non-high-grade serous ovarian cancer) and genitourinary cancers (urothelial cancer and clear cell renal cell carcinoma [ccRCC]).

DETAILED DESCRIPTION:
This trial is designed to evaluate the efficacy and safety of R-DXd in locally advanced or metastatic solid tumors with various CDH6 expression levels. Solid tumor types will include gynecological cancers (endometrial cancer, cervical cancer, and non-high-grade serous ovarian cancer) and genitourinary cancers (urothelial cancer and ccRCC).

For all cohorts except ccRCC, the primary endpoint will be objective response rate (ORR) by investigator assessment per RECIST 1.1. For the ccRCC cohort, the primary endpoint will be disease control rate (DCR) by investigator assessment per RECIST 1.1. All cohorts will also have the assessment of safety and tolerability as another primary objective.

ELIGIBILITY:
Participants must meet all of the following criteria to be eligible for enrollment into the trial:

1. Adults ≥18 years of age on the day of signing the ICF.
2. Participants must have at least 1 lesion, not previously irradiated, amenable to biopsy, and must consent to provide a pre-treatment biopsy from a primary and/or metastatic lesion.
3. Has at least 1 measurable lesion according to RECIST version 1.1 per investigator assessment.
4. Participants must have progressed radiologically on or after their most recent line of systemic therapy.
5. Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Additional inclusion criteria for endometrial cancer cohort

   1. Pathologically or cytologically documented endometrial cancer (carcinoma of any histological subtype or carcinosarcoma), irrespective of MSI or mismatch repair status.
   2. Documented disease progression after having received ≥1 line of therapy (no more than 3), including PBC-containing systemic treatment and an anti-PD-1 therapy containing regimen (combined or sequential) in the advanced/metastatic setting.
7. Additional inclusion criteria for cervical cancer cohort

   1. Pathologically or cytologically documented recurrent or persistent squamous, adenosquamous, or adenocarcinoma of the uterine cervix.
   2. Disease progression after having received ≥1 prior line of therapy that includes systemic therapy in the advanced or metastatic setting.
8. Additional inclusion criterion for non-HGSOC cohort

   a. Pathologically or cytologically documented unresectable or metastatic CCOC, low grade endometrioid, low-grade serous, or mucinous OVC that was previously treated with at least 1 prior line of therapy.
9. Additional inclusion criteria for urothelial cancer cohort

   1. Pathologically or cytologically documented unresectable or metastatic urothelial carcinoma of the bladder, renal pelvis, ureter, or urethra. Histological variants are allowed if urothelial histology is predominant.
   2. Relapsed or progressed after treatment with ≥1 prior line of therapy (maximum of 3) that contains anti-PD-(L)1 therapy in the perioperative or metastatic setting.
10. Additional inclusion criterion for the ccRCC cohort a. Pathologically or cytologically documented unresectable or metastatic ccRCC that was previously treated with no more than 3 prior systemic regimens for locally advanced or metastatic RCC, including both a PD-(L)1 checkpoint inhibitor and a VEGF-TKI in sequence or in combination.

Participants who meet any of the following criteria will be disqualified from entering the trial:

1. Clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis
2. Any of the following within the past 6 months prior to enrollment: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event.
3. Uncontrolled or significant cardiovascular disease as specified in the protocol.
4. Has a history of (noninfectious) ILD/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
5. Clinically severe pulmonary compromise
6. Chronic steroid treatment (>10 mg/day) with exceptions as noted in the protocol.
7. History of other active malignancy within 3 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (eg, 5-year OS rate >90%) and treated with expected curative outcome.
8. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE Version 5.0, Grade ≤1 or baseline.
9. Prior exposure to other CDH6-targeted agents or an ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan, datopotamab deruxtecan).
10. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection.
11. Has active or uncontrolled HIV, HBV, or HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate as Assessed by the Investigator (All Cohorts Except ccRCC) | Baseline up to 32 months
  Objective response rate (ORR) is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1 criteria.
Disease Control Rate (DCR) as Assessed by the Investigator (ccRCC Cohort Only) | Baseline up to 32 months
  Disease control rate (DCR) is defined as proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (maintained for ≥5 weeks) according to RECIST version 1.1.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) (All Cohorts) | Baseline up to 32 months

SECONDARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by the Investigator | Baseline up to 32 months
  Progression-free survival (PFS) is defined as the time interval from the start date of trial intervention to the date of radiographic disease progression according to RECIST version 1.1 criteria or death due to any cause, whichever comes first.
Duration of Response (DoR) as Assessed by the Investigator | Baseline up to 32 months
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (CR or PR) that is subsequently confirmed to the date of the first documentation of radiographic disease progression according to RECIST version 1.1 criteria or death due to any cause, whichever occurs first.
Time to Response (TTR) as Assessed by the Investigator | Baseline up to 32 months
  Time to response (TTR) is defined as the time from the start date of trial intervention to the date of the first documentation of response (CR or PR) that is subsequently confirmed. TTR will be calculated for confirmed responders only.
Objective Response Rate as Assessed by the Investigator (ccRCC Cohort Only) | Baseline up to 32 months
  Objective response rate (ORR) is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1 criteria.
Disease Control Rate (DCR) as Assessed by the Investigator (All Cohorts Except ccRCC Cohort) | Baseline up to 32 months
  Disease control rate (DCR) is defined as proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (maintained for ≥5 weeks) according to RECIST version 1.1.
Pharmacokinetic Parameter Maximum Concentration (Cmax) of R-DXd | Cycles 1 and 3 Day 1 predose and end of infusion (EOI), 3 hours (hr), and 5 hr postdose; Cycle 1 Days 8, 15, and 22; Cycle 2 Day 1 predose and EOI postdose; Cycle 4 (and every 2 cycles thereafter) predose, up to 32 months (each cycle is 21 days)
The Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive At Any Time and Who Have a Treatment-emergent ADA | Baseline up to 32 months

CONTACTS AND LOCATIONS:
Locations (48):
- United States (8):
  - Northside Hospital, Marietta, Georgia
  - University of Michigan Comprehensive Cancer Center Michigan Medicine, Ann Arbor, Michigan
  - Astera Cancer Care, East Brunswick, New Jersey
  - Women's Cancer Care Associates, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - West Cancer Center and Research Institute, Germantown, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - UZ Leuven Gynaec onco, Leuven
  - ZAS Sint-Augustinus, Wilrijk
- China (2):
  - Hunan Cancer Hospital, Changsha
  - Shanghai Cancer center, Shanghai
- Herlev og Gentofte Hosp, Copenhagen, Denmark
- France (9):
  - François Baclesse Center, Caen
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Grp Hsp Diac Croix Saint Simon, Paris
  - Cario - Centre Armoricain de Radiothérapie, Imagerie Médicale Et Oncologie, Plérin
  - Ico - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Italy (7):
  - AO per lEmergenza Cannizzaro, Catania
  - Irccs Ospedale San Martino, Genova
  - IRCCS Dino Amadori - IRST, Meldola
  - IRCCS San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Federico II Hospital, Naples
  - Azienda Ospedaliera S Maria, Terni
- Japan (8):
  - Hyogo Cancer Center, Akashi
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Aichi Cancer Centre, Nagoya
  - Osaka International Cancer Institute, Osaka
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Universitario de A Coruña, A Coruña
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital de Sant Pau, Barcelona
  - The Clínica Universidad de Navarra Madrid, Madrid
  - Md Anderson Cancer Centre, Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/